CLINICAL TRIAL: NCT00550511
Title: Randomized Study Evaluating the Role of Surgeon-Performed Ultrasound in the Management of the Acute Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ULABD-1
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Abdominal Pain
Keywords: Abdominal pain; ultrasound; surgery; emergency department; diagnostic accuracy
MeSH Terms: conditions — Abdominal Pain; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound (Other): Surgeon-performed ultrasound as intervention, as a complement to clinical investigation and standardized laboratory testing.
  Interventions: Radiation: Surgeon-performed ultrasound
- Control (No Intervention): Control group examined with clinical examination including standardized laboratory tests.

INTERVENTIONS:
Radiation: Surgeon-performed ultrasound — After clinical investigation including standardized laboratory tests the patient in the intervention arm is examined with abdominal ultrasound performed by the study surgeon.
  Other Names: US
  Arms: Ultrasound

SUMMARY:
The purpose of this study is to evaluate whether surgeon-performed ultrasound as a supplement to clinical investigation when a patient presents with abdominal pain in the emergency department can improve the management of the patient.

DETAILED DESCRIPTION:
Surgeon-performed ultrasound bedside in the emergency department when a patient presents with abdominal pain is quite common in Continental Europe and USA. It is considered to be implemented at emergency departments all over Sweden. This is the first randomized study performed to evaluate the method. In our study we compare diagnostic accuracy and further management of patients admitted to the emergency department for abdominal pain, with or without examination with surgeon-performed ultrasound bedside.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to emergency ward for abdominal pain
* 18 years or older

Exclusion Criteria:

* Pregnancy
* Condition that has to be taken care of immediately
* Inability to communicate with the investigator
* Previously diagnosed abdominal condition
* Severe drug or alcohol addiction
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2004-02; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Proportion of correct diagnosis | 6 weeks

SECONDARY OUTCOMES:
Time consumption in emergency department Time to decision about surgical intervention Amount of complementary examinations Amount of hospital admissions Patient satisfaction in the emergency ward and at follow up Consumption of health care | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Adami, ass prof, Principal Investigator — Karolinska Institutet, Department of Medicine, Clinical epidemiology unit; Anna Lindelius, MD, Study Director — Karolinska Institutet, Department of Surgery, Stockholm South General Hospital

REFERENCES:
- [Derived] Lindelius A, Torngren S, Nilsson L, Pettersson H, Adami J. Randomized clinical trial of bedside ultrasound among patients with abdominal pain in the emergency department: impact on patient satisfaction and health care consumption. Scand J Trauma Resusc Emerg Med. 2009 Nov 27;17:60. doi: 10.1186/1757-7241-17-60. PMID 19941671
- [Derived] Lindelius A, Torngren S, Pettersson H, Adami J. Role of surgeon-performed ultrasound on further management of patients with acute abdominal pain: a randomised controlled clinical trial. Emerg Med J. 2009 Aug;26(8):561-6. doi: 10.1136/emj.2008.062067. PMID 19625549